CLINICAL TRIAL: NCT01815983
Title: Does Video-Assisted Self Review Help Students Learn a New Skill Faster?
Brief Title: Video-Assisted Laryngoscopy Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 367729
Record Dates: First submitted 2013-03-07; First posted 2013-03-21 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Surgery
Keywords: Laryngoscopy; Tracheal Intubation; Video Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Videolaryngoscopy review. (Experimental): Video review.
  Interventions: Other: Videolaryngoscopy review.

INTERVENTIONS:
Other: Videolaryngoscopy review. — Review of video recordings.

SUMMARY:
This study is designed to evaluate the impact of a video recording review on the acquisition of a new technical skill (laryngoscopy and tracheal intubation).

ELIGIBILITY:
Inclusion Criteria:

* Medical students on elective rotation in anesthesiology.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Impact of videolaryngoscopy on skill acquisition. | 4 weeks
  Recorded intubations reviewed with volunteers learning a new skill.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Fleming, M.D., Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/study-to-examine-if-video-self-review-of-intubation-skills-by-medical-students-help-them-learn-the-skill-faster-851814/